CLINICAL TRIAL: NCT03600896
Title: Recombinant Human Interleukin-7 (CYT107) to Promote T-Cell Recovery After Cord Blood Transplantation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Supply issues from Sponsor
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Revimmune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0414; 2R01CA061508-21 (NIH); NCI-2018-01750 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Umbilical Cord Blood Transplant
Keywords: Umbilical Cord Blood Transplant; Recombinant human interleukin-7; CYT107; T-Cell Recovery after Cord Blood Transplantation; CBT
MeSH Terms: interventions — Interleukin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Recombinant Human Interleukin-7 (CYT107) (Experimental): In Part 1 of the study, 3 dose levels of CYT107 will be tested in this study. Up to 3 participants will be enrolled in each dose level. The first group of participants will receive the lowest dose level. The next group will receive a higher dose than the first group, if no intolerable side effects were seen. The third group will receive an even higher dose than the second, if no intolerable side effects were seen. Based on the results seen, 1 of the 3 doses will be selected as the recommended dose.
  In Part 2 of the study, an additional 25 participants will be enrolled to receive CYT107 at the recommended dose found in Part 1.
  Interventions: Drug: CYT107
- Phase 2: Recombinant Human Interleukin-7 (CYT107) (Experimental): In Part 2 of the study, an additional 25 participants will be enrolled to receive CYT107 at the recommended dose found in Part 1.
  Interventions: Drug: CYT107

INTERVENTIONS:
Drug: CYT107 — Phase I: Patients will be treated with CYT107 post CBT (from 60 to 180 days), in with 1 of 3 doses below:
  * 5 mcg/kg/dose for 3 doses
  * 10 mcg/kg/dose for 3 doses
  * 20 mcg/kg/dose for 3 doses
  The optimal recommended dose determined in Phase I will be used to treat all patient enrolled in Phase II.
  Other Names: Recombinant Human Interleukin-7

SUMMARY:
Participant is being asked to take part in this study because participant received an umbilical cord blood transplant as part of participant's standard treatment. Umbilical cord blood is a source of blood-forming cells that can be used for transplantation, also known as a graft.

The problem with this type of transplant is the small number of blood-forming cells available in cord blood transplants, which may delay the "take" of the graft in the transplant recipient.

There are 2 parts to this study.

The goal of Part 1 of this clinical research study is to learn if it is safe and practical to give recombinant human interleukin-7 (CYT107) to patients who have received a cord blood transplant. Researchers want to learn if CYT107 affects the "take" of the graft and the recovery of certain blood cells related to the immune system (called T-cells, NK cells, and B cells) in patients who have had a cord blood transplant.

The goal of Part 2 of this study is to learn if CYT107 may prevent or reduce the effects of graft-versus host disease (GVHD) or the likelihood of developing infections (such as cytomegalovirus [CMV], Epstein-Barr virus [EBV], and BK virus). GVHD happens when transplanted donor tissue attacks the tissues of the recipient's body.

This is an investigational study. CYT107 is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how CYT107 is designed to work.

Up to 34 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If participant is found to be eligible to take part in this study and participant agrees, participant will be assigned to a study group based on when participant joined this study.

In Part 1 of the study, 3 dose levels of CYT107 will be tested in this study. Up to 3 participants will be enrolled in each dose level. The first group of participants will receive the lowest dose level. The next group will receive a higher dose than the first group, if no intolerable side effects were seen. The third group will receive an even higher dose than the second, if no intolerable side effects were seen. Based on the results seen, 1 of the 3 doses will be selected as the recommended dose.

In Part 2 of the study, an additional 25 participants will be enrolled to receive CYT107 at the recommended dose found in Part 1.

Study Drug Administration:

Participant will be given one injection of CYT107 directly into the muscle 1 time each week for 3 weeks. If the doctor thinks it is needed, participant may be able to receive CYT107 as an injection under the skin instead of the muscle.

Participant will be given standard drugs to help decrease the risk of side effects. Participant may ask the study staff for information about how the drugs are given and their risks.

Length of Study Participation:

Participant may receive up to 3 injections of CYT107. Participant will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if participant is unable to follow study directions.

Participation in this study will be over about 1 year after the last injection.

Study Visits:

One (1) time each week during Weeks 1-3:

* Participant will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests.

Before each dose of CYT107 and then about 21, 28, and 100 days after the first injection, blood (about 1 tablespoon each time) will be drawn to check your immune system function, to check for infections, and to check the effects of CYT107 on participant's body.

One (1) time each week for about 6 months, blood (about 4 teaspoons) will be drawn to check for CMV. Part of the blood may be used to check for EBV. If participant has symptoms of BK infection during the study, blood (about 1 teaspoon) and urine will also be collected to check for the BK virus.

Pharmacokinetic (PK) and Research Testing:

Blood (about 1 tablespoon each time) will be drawn for PK testing before participant's first CYT107 injection and then 3 more times over the 24 hours after participant's first injection. Blood will also be drawn after participant's last CYT107 injection. PK testing measures the amount of study drug in the body at different time points.

Before the first CYT107 injection and on Day 42, blood (about 1 teaspoon each time) will be drawn to test for anti-CYT107 antibodies. Antibodies are created by the immune system and may attack foreign cells or substances, such as CYT107. If the test on Day 42 is positive, blood (about 1 teaspoon) will be drawn on Day 100 to check for CYT107 antibodies. These blood samples will be sent to the study supporter, Revimmune. After the samples are used for this antibody testing, the samples will be destroyed.

Follow-Up:

After participant's last dose of CYT107, participant will continue to have follow-up visits as part of participant's standard care (visits participant would have even if participant was not taking part in this study) for up to 1 year after participant's last dose. Information from these follow-up visits, such as results of any standard of care testing, will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years old or older.
2. Patient post a cord blood transplant (CBT) with documented absolute neutrophil engraftment and no evidence of GVHD or no history of acute or chronic GVHD requiring systemic steroids.
3. Patients with documented engraftment but require granulocyte colony-stimulating factor (G-CSF) for myelosuppressive antibiotics or antiviral medications are eligible.
4. Karnofsky performance status (KPS) > 60%.
5. Adequate organ function: Pulmonary: Absence of dyspnea or hypoxia (< 90% of saturation by pulse oximetry on room air).
6. Hepatic: Bilirubin </= 1.5 X ULN, AST (SGOT) and /or ALT (SGPT) </= 2.5 X ULN. PT/PTT < 1.5 X ULN.
7. Renal: Calculated Creatinine clearance > 60 mL/min/1.73 m2.
8. Diagnosis of acute myeloid leukemia; myelodysplastic syndrome; chronic myeloid leukemia or myeloproliferative disease.

Exclusion Criteria:

1. Pregnant or nursing.
2. History of lymphoid malignancy (including Hodgkin disease, non-Hodgkin lymphoma, Acute Lymphoblastic Leukemia and Chronic Lymphocytic Leukemia) or acute biphenotypic leukemia.
3. History of EBV associated lymphoproliferation.
4. Active uncontrolled viral, bacterial or fungal infection.
5. Documented human immunodeficiency virus (HIV)-1 or -2, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection at any time before or after transplant. (a positive hepatitis B serology indicative of a previous immunization is not an exclusion criteria).
6. EBV viremia equal to or greater than 500 copies EBV DNA/mL of blood by quantitative PCR.
7. History of autoimmune disease.
8. Receiving systemic corticosteroid therapy.
9. Receiving concurrent treatment with another investigational drug and/or biological agent.
10. Receiving anticoagulant therapy.
11. Uncontrolled hypertension.
12. QTc prolongation (QTc > 470 ms) or prior history of significant arrhythmia or ECG abnormalities.
13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
14. Any past or current psychiatric illness that, in the opinion of the investigator, would interfere with adherence to study requirements or the ability and willingness to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Toxicity of Recombinant Human Interleukin-7 (CYT107) defined as any of the events grade 3 or 4 GVHD, secondary graft failure, death, or grade 4 organ failure | Within 42 days of the first injection
Effects of Patient Covariates Variables on the Immune Reconstitution Parameters | Baseline up to 1 year post-IL-7
  Longitudinal Bayesian model used to assess the effects of patient covariates variables on the immune reconstitution parameters.
Rate of Viral Infections in CBT Patients Who Received Three Doses of CYT107 Following Engraftment | 3 weeks
  The observed rates of virus infections evaluated by tabulation and Bayesian regression modeling.

SECONDARY OUTCOMES:
Secondary Graft Failure | After CYT107 given up to one year
  Secondary graft failure defined as a sustained declined of ANC <0.5 x109/L for 3 consecutive days after initial documented engraftment with no evidence of disease progression.
Effects of Patient Treatment Variables on the Immune Reconstitution Parameters | Baseline up to 1 year post-IL-7
  Longitudinal Bayesian model used to assess the effects of patient treatment variables on the immune reconstitution parameters.

CONTACTS AND LOCATIONS:
Overall Officials: David Marin, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org